CLINICAL TRIAL: NCT04056078
Title: The Throwing Shoulder: The Cause of Shoulder Injuries or Pain in Experienced Handball Players: Nordic Throwing Shoulder Project (NTS - Project)
Brief Title: Nordic Throwing Shoulder Project (NTS - Project)
Status: Recruiting | Type: Observational
Sponsor: Nord University (Other)
Collaborators: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Tina Piil Torabi, PT, MSc. In Physical therapy and Sport Science, PhD. Student, Nord University
Other Study IDs: NordU
Record Dates: First submitted 2019-08-07; First posted 2019-08-14 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Shoulder Injuries; Shoulder Pain; Injury Prevention; Kinematics; Kinetics; Muscle Weakness; Throwing Performance; Overhead Injuries
MeSH Terms: conditions — Shoulder Injuries; Shoulder Pain; Muscle Weakness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Team Handball Players Playing with Shoulder Pain: Team Elite Handball players playing with shoulder pain i their dominated shoulder for more than 3 months.
- Team Handball Players playing without shoulder pain: Team Elite Handball players who never have experience shoulder pain i their dominated shoulder.
- Team Handball Players playing with previous shoulder pain: Team Handball players who have had shoulder pain i their dominated shoulder, but currently have been playing without shoulder pain in the previous 6 months.

SUMMARY:
As a part of the Olympic program and with 150 countries in the international Handball Federation team handball has become a worldwide popular sport. Unfortunately, a large number of different types injuries have been reported among team handball players, and shoulder pain has some of the biggest incidence. In handball 44-75% of the athletes had a history of shoulder pain and a weekly prevalence of shoulder problems in 28% of the athletes. Shoulder pain has been reported to have an impact on the athletes' training activities, performance, and daily life.

Several studies have established risk factors for shoulder injuries among overhead athletes, with a focus on the range of motion in glenohumeral joint (ROM), shoulder strength and scapula control. Injury occurrence results from a combination of possessing these different risk and the amount of throwing. Thereby training overhead sports must be considered a primary risk factor for shoulder injury.

However, several studies have performed kinematics analysis of different throws techniques commonly used in team handball. But no studies havn't investigated kinematics and kinetics of different throwing techniques in relation to team handball players and the development of shoulder pain, and if a throwing technique or a wrong throwing technique stresses the shoulder joint more than other throwing techniques. In baseball it was found that youth pitchers throwing with a curveball was associated with a 52% increased risk of shoulder pain and the slider was associated with an 86% increased risk of elbow pain, and there was a significant association between number of throws and rate of shoulder pain.

Two types of wind-ups are used in handball, and those different wind-ups also changed the throwing kinematics and throwing performance. Investigators found that the pelvis rotation was more important in the throw with the circular wind-up than in the whip-like wind up. In addition, the total throwing time was longer with the circular wind up. This could result in less stress and forces on the shoulder joint when compared with the whip like to reach the same performances.

The questions arises whether the used throwing techniques of the handball players during training and matches are a risk factor for shoulder pain and if some throwing techniques cause bigger risk than other throwing techniques as the players could put more force on the shoulder and elbow joint.

DETAILED DESCRIPTION:
For a trainer or a coach in sports, it is very important to know what determines performance and how to affect the performance by training. However, training can also cause injuries by using wrong techniques or too much overload. One of those injuries in handball (one of the biggest sports in Scandinavia) is shoulder pain. Besides handball, shoulder pain and injury is reported to be a large problem in athletes in other overhead sports such as baseball, javelin, tennis, badminton, volleyball. In handball 44-75% of the athletes had a history of shoulder pain and a weekly prevalence of shoulder problems in 28% of the athletes. While in baseball half of the youth baseball pitchers prevalence shoulder pain during the season. Shoulder pain has been reported to have an impact on the athletes' training activities, performance, and daily life.

Several studies have investigated risk factors for shoulder injuries among overhead athletes, with particular focus on glenohumeral joint range of motion (ROM) and shoulder strength. and scapular control.

In handball it was found that reduced glenohumeral internal rotation and excessive glenohumeral external rotation have been suggested as risk factors and that a reduction of total glenohumeral rotation has been associated with shoulder problems. Regarding rotator cuff strength, external rotation weakness and low ratios of concentric and eccentric external to internal rotation strength have been reported as risk factors in handball and baseball. In addition, weakness in glenohumeral abduction strength has been associated with shoulder injury in baseball. However, in a recent study of van Cingel the glenohumeral internal range of motion deficit and total range of motion deficit in elite female handball players seemed not to be risk factors for shoulder injuries.

However, sports injury research needs to move from simple analyses of risk factors and concentrate on how these factors interact among other determinants for injury. Athletes in overhead sports require a subtle balance of shoulder stability and mobility in order to meet the functional demands of their respective sport. It has been reported that altered shoulder mobility in these athletes is caused by adaptive structural changes to the joint because of the extreme physiological demands of the overhead activity. Nonetheless, it is not known if these possible changes that are necessary for high performance also cause injuries. Injury occurrence results from a combination of possessing these different risk factors and participating with these risk factors. Mostly it is a combination of possessing these risk factors and the amount of throwing that causes injuries. Thereby training overhead sports must be considered a primary risk factor for shoulder injury, while non-participation-related risk factors like strength, glenohumeral ROM and scapular control influence the amount of handball participation a player can tolerate before shoulder injury occurs. Møller showed in a 31-week cohort study of elite youth handball players that an increase in handball load by >60% was associated with greater shoulder injury rate. Furthermore, the effect of an increase in handball load between 20% and 60% was worsened among players with reduced external rotational strength or scapular dyskinesia.

However, none of the above mentioned studies investigated kinematics of throwing, which perhaps could be the most important risk factor for shoulder injuries.

A throwing technique or a wrong throwing technique that stresses the shoulder joint than other throwing techniques. In baseball it was found in youth pitchers that throwing with a curveball was associated with a 52% increased risk of shoulder pain and the slider was associated with an 86% increased risk of elbow pain. There was a significant association between the number of pitches thrown in a game and during the season and the rate of elbow pain and shoulder pain. The investigators concluded that pitchers in this age group should be cautioned about throwing breaking pitches (curveballs and sliders) because of the increased risk of elbow and shoulder pain and that a limitation on pitches thrown in a game and in a season can reduce the risk of pain. In another study showed other risk factors like decreased satisfaction, arm fatigue during the game pitched, throwing more than 75 pitches in a game, and throwing fewer than 300 pitches during the season.

In handball, it is difficult to count all throws during training and matches. However, it is possible to perform kinetic and kinematic and neuromuscular analysis of these types of throws. Several studies have performed kinematics analysis of different throws in handball. In these studies kinematics of different types of throws like standing, with run up and jump throws, which are the three commonly used types of throws in team handball were analyzed.

It was shown that the elbow extension and internal rotation movement starting from a maximal external rotation angle is one of the main contributors in overarm throwing in team handball. Furthermore it was thought that hypermobility (increased maximal external rotation angle) in the overhead athletes to allow larger arm cocking might have a positive effect on ball velocity.

Yet, this mobility of the overhead athletes is often tested by active and passive range of motion tests conducted by physical therapists. In these tests the maximal glenohumeral internal and external rotation angle is measured and used as a measurement of shoulder mobility. Furthermore, the range of motion of the glenohumeral joint is compared with a normal population or with the non-dominant arm. In addition, most studies that conducted these types of measurements were performed in baseball and tennis. As described earlier changes in the range of motion measured during these tests were identified as risk factors. Still, none of these studies have investigated whether the measured range of motion of the external rotation also influences the actual throwing kinematics. Only one study reported in baseball players that there was a correlation between passive range of motion of external rotation and the maximal external rotation angle during pitching. On the other hand, in handball a study did not find any correlation between these ROM tests and throwing kinematics or performance in elite team handball throwers.

The questions arises whether the used throwing techniques of the handball players during training and matches are a risk factor for shoulder pain and if some throwing techniques cause bigger risk than other throwing techniques as it could put more force on the shoulder and elbow joint.

A study identified that all used handball throws can be divided by their wind-up: a circular or whip-like wind up and that these different wind up cause different important changes in the throwing kinematics and throwing performance. The investigators found that the pelvis rotation was more important in the throw with the circular wind-up than in the whip-like wind up. In addition, the total throwing time was longer with the circular wind up. This could result in less stress and forces on the shoulder joint when compared with the whip like to reach the same performances. However, only standing throws were investigated and no kinetic analysis (inverse dynamics) were performed that could show how much force there occurs upon the shoulder joint during different throws. Furthermore, to the best of our knowledge, also no neuromuscular investigations of the muscles used during the different handball throwing techniques are performed to give more insight about the muscle use during handball throws that produce the different joint movements and have to manage the kinetics on the shoulder joint.

Following research questions are expected answered during this project.

1. How do the three most used techniques in team handball (standing, with run-up and jump throws), with different wind-ups (circular and whip-like) influence the kinematics, the neuromuscular coordination and kinetics in the shoulder joint (anterior and posterior peak force)?
2. Do previous shoulder injury/pain, current injury/pain or post- shoulder operation influence on the throwing biomechanics and neuromuscular coordination compared with handball players playing without pain?
3. How do shoulder strength, stability and trunk mobility influence throwing kinematics and kinetics?

ELIGIBILITY:
Inclusion Criteria:

* Elite handball players in the top three leagues in Denmark, Sweden and Norway
* Players playing without shoulder pain.
* Players playing with previous shoulder.
* Players playing with shoulder pain.
* Participating in both defends- and attack- relating situations.

Exclusion Criteria:

* Operation in the shoulder
* Not participating in attack related situations.
* Shoulder pain caused by a traumatic event

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Elite Team Handball players playing in the top 3 leauges in Scandinavia will be invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-02-24 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-02 (Estimated)

PRIMARY OUTCOMES:
The change of joint positions and joint movements in the shoulder during overhead throws | Day 1
  Kinematic (joint movement) of the upperbody during different styles overhead throws. Ball velocity and throwing kinematics will be measured using a 3D motion capture system (Qualysis, Sävedalen, Sweden, eight cameras, 240-500 Hz) tracking the position of the reflective markers (2.6 cm diameter) during the hole movement.
Generated joint forcers in the shoulder during overhead throws | Day 1
  Joint forces (Kinetics) will be measured by using a 3D motion capture system (Qualysis, Sävedalen, Sweden, eight cameras, 240-500 Hz) and calculated by the theory of inverse dynamics of the upperbody during different styles of overhead throws. Kinetics measured by inverse dynamics will be calculated with Visual 3D (C-Motion, Germantown, MD) or Simi motion systems, and the forces in the shoulder will be presented in Newton.
Upperbody Muscle Activity during different styles overhead throws | Day 1
  Muscular activity will be measured by electromyography (EMG). Muscles relevant to investigate the throwing technique will be measured with Bipolar surface EMG electrodes.

SECONDARY OUTCOMES:
Scapula-humeral Control | Day 1
  Scapula Control will be measured using the scapula dyskinese test (SDT).
Range of Motion | Day 1
  The passive range of glenohumeral Internal Rotation and External Rotation will be measured using a electric goniometer.
Strength | Day 1
  Isometric strength in the glenohumeral Internal Rotation and External rotation muscles will be measured using a handheld dynamometer.
Shoulder and trunk stability | Day 1
  CKCUES test will be used to the ability to resist an external standardized perturbation
Oslo Sports Trauma Reseach Center Overuse Injury Questionnaire | Day 1
  The questionnaire will be used to measure shoulder pain and injury registration among elite handball players.
  The OSTRC include 4 questions regarding; Difficulties in participating, Reduced training volumne, Affected performance and pain related to their sport. Each question must be answered by the presented 4-5 categories.
  Each category is allocated with a numerical value from 0 to 25, and these are summed in order to calculate a servity score from 0 to 100 for each problem.
WOSI questionnaire | Day 1
  The questionnaire will be used to measure shoulder pain and injury registration among elite handball players.
  WOSI includes in total 21 questions, which is devided in 4 subcategories; Physical Symptoms question 1-10, Sports/recreation/work question 11-14, Lifestyle question 15-18 and Emotion question 19-21.
  A total score varies from 0 point - to maximal of 2100 point.

CONTACTS AND LOCATIONS:
Locations (2):
- Human Movement Laboratory, Hvidovre Hospital, Hvidovre, København, Denmark
- Nord University, Levanger, Norway

IPD SHARING:
Plan to Share IPD: Undecided
We havn't decided whether the data should be shared by other researchers.